CLINICAL TRIAL: NCT05857358
Title: Safety and Potential Effect of Innovative Cell-based Therapy Using Adipose-derived Stromal Vascular Fraction in Patients With Autoimmune Xerostomia (XEROCELL)
Brief Title: Safety and Potential Effect of Innovative Cell-based Therapy Using Adipose-derived Stromal Vascular Fraction in Patients With Autoimmune Xerostomia
Acronym: XEROCELL
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-505149-20-00
Record Dates: First submitted 2023-04-14; First posted 2023-05-12 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Xerostomia
MeSH Terms: conditions — Xerostomia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adult patients suffering from xerostomia and autoimmune disease (Experimental): Xerostomia treatment consist of 3 steps (including 2 surgical steps) in the Hospital de la Conception of Marseille, in the same ward :
  * The plastic/maxillofacial surgeon : collects the adipose tissue, and transfers it to the cell therapy unit;
  * The cell therapy unit processes and controls the experimental product (adipose-derived stromal vascular fraction; AD-SVF) from the harvested adipose tissue. The AD-SVF batch is nominatively transported to the surgeon;
  * The maxillofacial surgeon injects the AD-SVF without delay under local anesthesia.
  Interventions: Procedure: lipoaspiration; Drug: Injection of the autologous adipose-derived stromal vascular fraction (AD-SVF)

INTERVENTIONS:
Procedure: lipoaspiration — Adipose tissue harvest will be conducted by a surgeon under under local and intra-veinous sedation anesthesia. Once the patient is asleep and just before the laying of the operating drapes, the skin will be thoroughly disinfected, in order to avoid bacteriological contamination. Each entry point will be disinfected with betadine before and regularly during the procedure and will receive local anesthesia.
  The lipoaspiration sites will be infiltrated using a closed system, thanks to a Khoury canula. Adipose tissue will be harvested after waiting at least 5 minutes, in order to limit hematoma and excessive blood harvesting. A 3mm incision will be made then the tissue collection will be performed using a canula, manually, by gentle aspirations into a syringe then directly transferred into a connected sterile bag.
  The incision will be closed with 1 stitch of 6-0 absorbable and a paraffin gauze dressing. Then, patient will be awaken and transported to the recovery room.
Drug: Injection of the autologous adipose-derived stromal vascular fraction (AD-SVF) — Autologous uncultured (AD-SVF) will be isolated by digestion and centrifugation of adipose tissue from lipoaspiration.
  Then, AD-SVF will be injected in 6 sites :
  * 2 for the accessory labial glands (0.5mL in the upper lip and 0.5mL in the lower lip)
  * 2 for the sublingual glands (0.5mL for each gland)
  * 2 for the inner face of cheeks (0.5mL for each side)
  The volume of injection will be of 3 mL containing 30 millions of AD-SVF viable nucleated cells for the total safety dose.

SUMMARY:
The main objective of this study is to evaluate the tolerance and safety of autologous adipose-derived stromal vascular fraction injected in accessory salivary glands for treatment of autoimmune xerostomia in terms of adverse reactions through day 14 (D14).

DETAILED DESCRIPTION:
Autoimmune xerostomia is a disabling condition affecting mostly patients suffering from Sjögren's disease, systemic lupus erythematosus, rheumatoid arthritis and systemic xerostomia.

Local therapies and systemic drug treatments (picarpine) remain the gold standards but have limited effects upon salivary flow action and many adverse effects.

Stem cell therapies and notably adipose tissue-derived stromal cells have shown promising potential for tissue repair. Autologous uncultured adipose-derived stromal vascular fraction (AD-SVF) is recognized as an easily accessible (by a standard lipoaspiration to obtain adipose tissue, from which AD-SVF are isolated by centrifugation), safe and well tolerated source of cells with angiogenic, anti-inflammatory, immunomodulatory and regenerative properties.

The purpose of our AD-SVF phase I trial is to evaluate, first the tolerance of autologous AD-SVF cells locally injected in the oral cavity and second their capability to improve the salivary function.

ELIGIBILITY:
Inclusion Criteria:

* Patients from 18 to 65 years.
* Patients suffering from xerostomia and autoimmune disease including : Gougerot-Sjögren disease according to AC/EULAR criteria and Secondary Gougerot-Sjögren syndrome related to systemic diseases (sclerodermia, rheumatoid arthritis, systemic lupus erythematosus...)
* Xerostomia visual scale (6-item visual analogue scale questionnaire) for assessment of salivary dysfunction : score ≥ 30/60
* Informed consent to participate (with signature)
* Negative β -HCG test and effective contraception for women being able to get pregnant
* Affiliation to the social security system

Exclusion Criteria:

* Medical history of head and neck neoplasia
* Recent (<3 months) medication inducing and aggravating xerostomia : Standard treatment with tricyclic antidepressant and/or antipsychotics
* Body Mass Index < 18
* Active smoking (> 5 cigarettes a day)
* Active infectious disease and/or active viral serologies (HIV, HCV, HBV, HTLV I/II, TPHA/VDRL)
* Coagulation disorders including anticoagulant and antiplatelet treatment
* Any temporary or definitive contraindication due to any medical or surgical unstable condition
* Allergy to local anesthesia and/or albumin
* Pregnant or breastfeeding women
* Adult protected by the law (tutorship and curatorship)
* Patients already enrolled in another study
* Patients under 18 years of age
* Person deprived of liberty
* Patient non-affiliated to the social security

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Intensity of adverse reactions at the injection site at day 1 | 1 day
  1 day after ADSVF injection, a subjective evaluation will be done by the patient of lip sensibility, pain, oedema or ecchymosis bleeding or haematoma, bleeding or haematoma, other event through an adapted report form with phone assessment
Intensity of adverse reactions at the injection site at day 3 | 3 days
  3 days after ADSVF injection, a subjective evaluation will be done by the patient of lip sensibility, pain, oedema or ecchymosis bleeding or haematoma, bleeding or haematoma, other event through an adapted report form with phone assessment.
Intensity of adverse reactions at the injection site at day 7 | 7 days
  7 days after ADSVF injection, a subjective evaluation will be done by the patient of lip sensibility, pain, oedema or ecchymosis bleeding or haematoma, bleeding or haematoma, other event through an adapted report form with clinical assessment.
Intensity of adverse reactions at the injection site at day 14 | 14 days
  14 days after ADSVF injection, a subjective evaluation will be done by the patient of lip sensibility, pain, oedema or ecchymosis bleeding or haematoma, bleeding or haematoma, other event through an adapted report form with clinical assessment.
Intensity of adverse reactions at the harvesting site at day 1 | 1 day
  1 day after ADSVF injection, a subjective evaluation will be done by the patient of pain, oedema or ecchymosis bleeding or haematoma, inflammation or infection, other event through an adapted report form with phone assessment.
Intensity of adverse reactions at the harvesting site at day 3 | 3 days
  3 days after ADSVF injection, a subjective evaluation will be done by the patient of pain, oedema or ecchymosis bleeding or haematoma, inflammation or infection, other event, through an adapted report form with phone assessment.
Intensity of adverse reactions at the harvesting site at day 7 | 7 days
  7 days after ADSVF injection, a subjective evaluation will be done by the patient of pain, oedema or ecchymosis bleeding or haematoma, inflammation or infection, other event, through an adapted report form with clinical assessment.
Intensity of adverse reactions at the harvesting site at day 14 | 14 days
  14 days after ADSVF injection, a subjective evaluation will be done by the patient of pain, oedema or ecchymosis bleeding or haematoma, inflammation or infection, other event through an adapted report form with clinical assessment.

SECONDARY OUTCOMES:
Intensity of adverse reactions at the injection site at day 15 | 15 days
  15 days after ADSVF injection, a subjective evaluation will be done by the patient of lip sensibility, pain, oedema or ecchymosis bleeding or haematoma, bleeding or haematoma, other event through an adapted report form with clinical assessment.
Intensity of adverse reactions at the injection site at month 1 | 1 month
  1 month after ADSVF injection, a subjective evaluation will be done by the patient of lip sensibility, pain, oedema or ecchymosis bleeding or haematoma, bleeding or haematoma, other event through an adapted report form with clinical assessment.
Intensity of adverse reactions at the injection site at month 3 | 3 months
  3 months after ADSVF injection, a subjective evaluation will be done by the patient of lip sensibility, pain, oedema or ecchymosis bleeding or haematoma, bleeding or haematoma, other event through an adapted report form with clinical assessment.
Intensity of adverse reactions at the injection site at month 6 | 6 months
  6 months after ADSVF injection, a subjective evaluation will be done by the patient of lip sensibility, pain, oedema or ecchymosis bleeding or haematoma, bleeding or haematoma, other event through an adapted report form with clinical assessment.
Intensity of adverse reactions at the injection site at month 7 | 7 months
  7 months after ADSVF injection, a subjective evaluation will be done by the patient of lip sensibility, pain, oedema or ecchymosis bleeding or haematoma, bleeding or haematoma, other event through an adapted report form with clinical assessment.
Intensity of adverse reactions at the harvesting site at day 15 | 15 days
  15 days after ADSVF injection, a subjective evaluation will be done by the patient of pain, oedema or ecchymosis bleeding or haematoma, inflammation or infection, other event through an adapted report form with clinical assessment.
Intensity of adverse reactions at the harvesting site at month 1 | 1 month
  1 month after ADSVF injection, a subjective evaluation will be done by the patient of pain, oedema or ecchymosis bleeding or haematoma, inflammation or infection, other event through an adapted report form with clinical assessment.
Intensity of adverse reactions at the harvesting site at month 3 | 3 months
  3 months after ADSVF injection, a subjective evaluation will be done by the patient of pain, oedema or ecchymosis bleeding or haematoma, inflammation or infection, other event through an adapted report form with clinical assessment.
Intensity of adverse reactions at the harvesting site at month 6 | 6 months
  6 months after ADSVF injection, a subjective evaluation will be done by the patient of pain, oedema or ecchymosis bleeding or haematoma, inflammation or infection, other event through an adapted report form with clinical assessment.
Intensity of adverse reactions at the harvesting site at month 7 | 7 months
  7 months after ADSVF injection, a subjective evaluation will be done by the patient of pain, oedema or ecchymosis bleeding or haematoma, inflammation or infection, other event through an adapted report form with clinical assessment.
primary efficiency of AD-SVF iin term of glands reparation process/repair (Minor salivary gland biopsy) | 6 months
  A minor salivary gland biopsy will be done under local anaesthesia 6 months after the injection. Then, an Histological analysis (4 grades Chilson-Mason score) of minor salivary gland biopsy will be performed.
efficacy of AD-SVF at month 1 | 1 month
  Salivary flow will be collected after stimulation 1 month after the injection. It is expressed in milliliter by minutes after 5 minutes of collect, and oligoptyalism isdefined by a salivary flow < 0.1 mL/mn at rest, and < 0.7 ml/mn after stimulation.
efficacy of AD-SVF at month 3 | 3 months
  Salivary flow will be collected after stimulation 3 months after the injection. It is expressed in milliliter by minutes after 5 minutes of collect, and oligoptyalism isdefined by a salivary flow < 0.1 mL/mn at rest, and < 0.7 ml/mn after stimulation.
efficacy of AD-SVF at month 6 | 6 months
  Salivary flow will be collected after stimulation 6 months after the injection. It is expressed in milliliter by minutes after 5 minutes of collect, and oligoptyalism isdefined by a salivary flow < 0.1 mL/mn at rest, and < 0.7 ml/mn after stimulation.
Change in dryness of oral mucosa | 3 months
  Change in dryness of oral mucosa will be assessed from Clinical Oral Dryness Score (CODS) based on 10 items realized before and, 3 and 6 months after the injection.
Change in xerostomia Visual Analogic Scale (VAS) | 6 months
  Change in VAS will be assessed from a 6-items questionnaire scored from 0 to 10 (increasing gravity) according to Likert scale.

IPD SHARING:
Plan to Share IPD: No